CLINICAL TRIAL: NCT06606873
Title: Anatomical Risk Factors for Orbital Complications in Patients With Acute Rhinosinusitis
Brief Title: Complicated Rhinosinusitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Abd El_Atty Sayed Harb, Doctor, Assiut University
Other Study IDs: Orbital complications of AR
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Orbital Complications of Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rhinosinusitis is among the most common conditions encountered in the primary care clinic.

DETAILED DESCRIPTION:
serious sequelae of ARS, including orbital and intracranial complications as Like Periorbital oedema and Displaced globe and Double vision and Ophthalmoplegia Reduced visual acuity

ELIGIBILITY:
Inclusion Criteria:

* Patients with orbital complications of rhinosinusitis

Exclusion Criteria:

* 1- Previous maxillofacial trauma history. 2- Previous nasal or paranasal surgery. 3- Invasive fungal rhinosinusitis. 4- Cases with odontogenic rhinosinusitis. 5- Immotile cilia syndrome, cystic fibrosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OBSERVATIONAL Split-half case-comparison study.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Orbital complications of rhinosinusitis | One year
  The presence of agger nasi cells (AGC), concha bullosa, Haller, Onodi or frontal recess cells, septal deviation, lower turbinate hypertrophy and hypoplasia or agenesis of the PNS

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelaziz, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lucas JW, Schiller JS, Benson V. Summary health statistics for U.S. adults: National Health Interview Survey, 2001. Vital Health Stat 10. 2004 Jan;(218):1-134. PMID 15791758
- [Result] Mekhitarian Neto L, Pignatari S, Mitsuda S, Fava AS, Stamm A. Acute sinusitis in children: a retrospective study of orbital complications. Braz J Otorhinolaryngol. 2007 Jan-Feb;73(1):75-9. doi: 10.1016/s1808-8694(15)31126-5. PMID 17505603
- [Result] Sedaghat AR, Wilke CO, Cunningham MJ, Ishman SL. Socioeconomic disparities in the presentation of acute bacterial sinusitis complications in children. Laryngoscope. 2014 Jul;124(7):1700-6. doi: 10.1002/lary.24492. Epub 2013 Dec 11. PMID 24338779